CLINICAL TRIAL: NCT02490319
Title: Study on the Biological Prediction Models of Radiation Pneumonitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianglin Yuan, Professor, Chief Physician, Huazhong University of Science and Technology
Other Study IDs: TJCC002
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Radiation Pneumonitis
Keywords: radiation pneumonitis; lung cancer; prediction models; genetic variants
MeSH Terms: conditions — Radiation Pneumonitis; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — From peripheral blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Lung cancer patients treated with thoracic radiation therapy

SUMMARY:
Radiation pneumonitis is the most common complication and the major dose-limiting toxicity associated with radiotherapy, which can cause poor quality of life or life-threatening symptoms and might hinder the tumor-controlling effects of radiotherapy. Consequently, establishing reliable predictors for the occurrence of RP is of great significance such that the therapeutic effects of RT can be maximized while minimizing its adverse effects. The aim of this study is to figure out the biological prediction models of radiation pneumonitis.

DETAILED DESCRIPTION:
1. Establish a clinical data base for the lung cancer patients treated with radiotherapy in Tongji Hospital.

   Data including age, gender, smoking state, KPS, pulmonary function, disease history, histology, stage, surgery, chemotherapy, dosimetric parameters of radiotherapy were collected.

   Peripheral blood was collected from all patients enrolled. All patients enrolled in this study are examined during and one month after radiotherapy. Then, the patients are followed every three months for the first year and every six months thereafter. At each follow-up visits, all patients are asked to undergo a chest X-ray or CT and clinical information, including symptoms, is collected. RP is graded by two radiation oncologists according to the Common Terminology Criteria for Adverse Events 4.0.
2. Select candidate genes and pathways which may be associated with radiation pneumonitis and identify their tagSNPs by Haploview.
3. Use Kaplan-Meier and Cox model to analyze the association of all the factors collected with radiation pneumonitis.
4. Establish a biological prediction models for radiation pneumonitis based on the statistics analysis

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of lung cancer by histology
2. Radiation dose at least 45 Gy
3. KPS>60
4. Life expectancy of at least 6 months
5. Voluntarily signed the informed consent

Exclusion Criteria:

1. Previous thoracic irradiation
2. Severe cardiopulmonary diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients treated with radiation therapy at Tongji Hospital, Huazhong University of Science and Technology (Wuhan, Hubei Province, China).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-09; Primary Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
radiation pneumonitis grade >=2 or 3 | 12 months after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Xianglin Yuan, MD, PhD, Principal Investigator — Tongji Hospital
Locations (1):
- Department of Oncology, Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Background] Mehta V. Radiation pneumonitis and pulmonary fibrosis in non-small-cell lung cancer: pulmonary function, prediction, and prevention. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):5-24. doi: 10.1016/j.ijrobp.2005.03.047. PMID 15963660
- [Background] Marks LB, Bentzen SM, Deasy JO, Kong FM, Bradley JD, Vogelius IS, El Naqa I, Hubbs JL, Lebesque JV, Timmerman RD, Martel MK, Jackson A. Radiation dose-volume effects in the lung. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S70-6. doi: 10.1016/j.ijrobp.2009.06.091. PMID 20171521
- [Background] Yuan X, Liao Z, Liu Z, Wang LE, Tucker SL, Mao L, Wang XS, Martel M, Komaki R, Cox JD, Milas L, Wei Q. Single nucleotide polymorphism at rs1982073:T869C of the TGFbeta 1 gene is associated with the risk of radiation pneumonitis in patients with non-small-cell lung cancer treated with definitive radiotherapy. J Clin Oncol. 2009 Jul 10;27(20):3370-8. doi: 10.1200/JCO.2008.20.6763. Epub 2009 Apr 20. PMID 19380441
- [Derived] Tang Y, Yang L, Qin W, Yi MX, Liu B, Yuan X. Impact of genetic variant of HIPK2 on the risk of severe radiation pneumonitis in lung cancer patients treated with radiation therapy. Radiat Oncol. 2020 Jan 8;15(1):9. doi: 10.1186/s13014-019-1456-0. PMID 31915028
- [Derived] Tang Y, Yang L, Qin W, Yi M, Liu B, Yuan X. Validation study of the association between genetic variant of IL4 and severe radiation pneumonitis in lung cancer patients treated with radiation therapy. Radiother Oncol. 2019 Dec;141:86-94. doi: 10.1016/j.radonc.2019.09.002. Epub 2019 Sep 17. PMID 31540745
- [Derived] Tang Y, Liu B, Li J, Wu H, Yang J, Zhou X, Yi M, Li Q, Yu S, Yuan X. Genetic variants in PI3K/AKT pathway are associated with severe radiation pneumonitis in lung cancer patients treated with radiation therapy. Cancer Med. 2016 Jan;5(1):24-32. doi: 10.1002/cam4.564. Epub 2015 Dec 8. PMID 26645682